CLINICAL TRIAL: NCT05384925
Title: Prior Abdominal Surgery: A Potential Risk Factor for Colonic Diverticulosis or Diverticulitis
Status: Completed | Type: Observational
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Principal Investigator, Eran Ariam, principal investigator, Assaf-Harofeh Medical Center
Other Study IDs: 0107-20
Record Dates: First submitted 2022-05-12; First posted 2022-05-20 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Diverticulosis, Colonic; Abdominal Adhesion; Diverticulitis
MeSH Terms: conditions — Diverticulosis, Colonic; Diverticulitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: comparison — abdominal surgery as a risk factor for diverticulosis

SUMMARY:
Background & Aims:

Abnormal colonic pressure profiles have been associated with an increased risk of colonic diverticulosis. A surgical history is a known risk factor for abdominal adhesions, and these may lead to increased intraluminal colonic pressure. We assessed whether previous abdominal surgery is associated with colonic diverticulosis or diverticulitis.

Methods:

The investigators analyzed data from a prospective study of patients undergoing colonoscopy for different indications from 2020 through 2021. Patients completed a structured questionnaire concerning previous abdominal surgeries, dietary and lifestyle exposures including smoking and alcohol use, and co-morbidities.

ELIGIBILITY:
Inclusion Criteria:

* patients > 18 years old who are going through colonoscopy in shamir medical center for any reason

Exclusion Criteria:

* inadequate preparation (Boston Bowel Preparation Quality Scale <6);
* previous colonic resection based on history and colonoscopy;
* previous colon cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients 18 years of age and older presenting for a colonoscopy at Shamir Medical Center between 2020 and 2021
Sampling Method: Probability Sample
Enrollment: 359 (Actual)
Dates: Start 2020-04-12 (Actual); Primary Completion 2021-05-22 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
correlation between prior abdominal surgery and the development of diverticulosis | in the end of the study (estimated in 1 year)
  the investigators are willing to see if prior abdominal surgery raise the patient's risk of developing future diverticulosis. The investigators use questionere to collect data from patients. The final measurements will be calculatrd with spss software

CONTACTS AND LOCATIONS:
Locations (1):
- Asag Harofeh Medical Center, Be’er Ya‘aqov, Israel

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code